CLINICAL TRIAL: NCT03293654
Title: A Randomised, Double Blind, Three-Arm, Single Dose, Parallel Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02 (Bevacizumab Biosimilar Drug), US Licenced Avastin® and EU Approved Avastin® in Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing MB02 And US And EU Avastin® In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB02 A 02 17
Record Dates: First submitted 2017-09-13; First posted 2017-09-26 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB02 (Bevacizumab Biosimilar) (Experimental): Intervention Description: Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: MB02
- US licenced Avastin® (Active Comparator): Intervention Description: Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: US licenced Avastin®
- EU approved Avastin® (Active Comparator): Intervention Description: Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: EU approved Avastin®

INTERVENTIONS:
Drug: MB02 — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion.
  Other Names: MB02 (Bevacizumab Biosimilar)
  Arms: MB02 (Bevacizumab Biosimilar)
Drug: US licenced Avastin® — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion.
  Other Names: Bevacizumab (United States)
  Arms: US licenced Avastin®
Drug: EU approved Avastin® — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion.
  Other Names: Bevacizumab (European Union)
  Arms: EU approved Avastin®

SUMMARY:
Randomized, double blind, parallel group, single dose, 3 arm study to investigate and compare the Pharmacokinetics (PK), safety and immunogenicity profile of MB02 with US and EU Avastin® in healthy male subjects.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary PK parameters are Cmax and AUC(0-∞). The PK parameters for bevacizumab will be calculated using standard noncompartmental methods. An analysis of covariance model will be used to analyse the log-transformed primary PK parameters (AUC[0-∞].and Cmax) and AUC(0-t). The model will include a fixed effect for treatment and body weight as a covariate.

All other PK parameters will not be subject to inferential statistical analysis. Estimates of geometric mean ratios together with the corresponding 90% confidence intervals will be derived for the comparisons of the PK parameters as follows:

* MB02 versus EU Avastin®
* MB02 versus US Avastin®
* EU Avastin® versus US Avastin®

PK similarity will be achieved if the 90% confidence intervals (CIs) for the biosimilar-to-reference ratios of PK endpoints (AUC[0-∞] and Cmax) fall within the predefined 0.80-1.25 acceptance similarity criteria for all 3 pairwise comparisons; MB02 versus EU-approved Avastin®; MB02 versus US-licenced Avastin®; and EU-approved Avastin® versus US-licenced Avastin®.

All AEs will be listed and summarised using descriptive methodology. All observed or patient-reported AEs will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. The incidence of AEs for each treatment will be presented by severity and by association with the study drugs as determined by the Investigator (or designee). All safety data will be listed and summarised as appropriate

Immunogenicity data (overall anti-drug antibody [ADA] incidence and titers, and neutralising ADA results) will be listed. A summary of the number and percent of subjects testing positive for ADA or neutralising antibodies before the dose of MB02, EU Avastin®, or US Avastin® (Day 1) and at scheduled postdose assessments will be presented by treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any race, between 18 and 55 years of age, inclusive, at Screening.
2. Body mass index between 18.5 and 29.9 kg/m2, inclusive, at Screening.
3. Total body weight between 60 and 95 kg, inclusive, at Screening.
4. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
5. Relevant clinical laboratory evaluations of haematology, coagulation, urinalysis and clinical chemistry within normal range at Screening and Check in as follows. A single repeat test will be allowed at each timepoint.

   * Absolute neutrophil count ≥1.5 × 109 L
   * Platelet count ≥100 × 109 L
   * Haemoglobin >10 g/dl
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN
   * Alkaline phosphatase (ALP) ≤1.5 × ULN
   * Total bilirubin <1.5 × ULN (<51.30 µmol/L in subjects with Gilbert's syndrome)
   * Blood urea nitrogen ≤1.5 × ULN
   * Creatinine < 132.63 µmol/L
   * Serum albumin: >35 g/L
   * Low density lipoprotein cholesterol ≤ ULN
   * High density lipoprotein cholesterol ≥ lower limit of normal
   * Creatine kinase (CK) < × 2 ULN
   * International normalised ratio (INR) 0.8-1.3
   * Urine dipstick for proteinuria <2+
6. Systolic blood pressure ≥90 mmHg and ≤140 mmHg and diastolic blood pressure ≥50 mmHg and ≤90 mmHg at Screening and Check in.
7. Subjects agree to use contraception as detailed in protocol.
8. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions. Subjects must have signed an informed consent before any study-related procedure or evaluation is performed.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Any current or recent history of active infections, including localised infections.
4. History of, or planned surgery, including suturing, dental surgery or wound dehiscence within 30 days of dosing, or within 30 days of the last study visit.
5. Presence of a nonhealing wound or fracture.
6. Known history of clinically significant essential hypertension, orthostatic hypotension, fainting spells or blackouts for any reason, cardiac failure or history of thromboembolic conditions.
7. Medically significant dental disease or dental neglect, with signs and/or symptoms of local or systemic infection that would likely require a dental procedure during the course of the study.
8. Clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to Check-in, and/or positive alcohol breath test and/or urinary drug test screen at Screening or Check in.
9. History of bleeding disorders or protein C, protein S, and/or factor V Leiden deficiency.
10. History of clinically signifiant haemorrhage, epistaxis, GI bleeding, haemorrhoids and/or haemoptysis.
11. History of GI perforation, ulcers, gastro oesophageal reflux, inflammatory bowel disease, diverticular disease, or any fistulae.
12. Alcohol consumption of >24 units per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
13. Positive hepatitis panel, positive human immunodeficiency test. Subjects whose results are compatible with prior immunisation and not infection may be included at the discretion of the Investigator.
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to Check-in, or within 5 half lives of the investigational drug used in the study.
15. Use or intend to use slow-release medications/products considered to still be active within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
16. Use or intend use of any prescription medications/ nonprescription products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator or designee.
17. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
18. Have received a live or attenuated vaccine from 3 months prior to Screening, or have the intention to receive a vaccine during the study.
19. Intend to travel to a region where a vaccination will be required due to endemic disease within 3 months of dosing.
20. Previous treatment with an anti VEGF antibody or any other protein or antibody targeting the VEGF receptor.
21. Use of tobacco- or nicotine-containing products within 5 years prior to Check-in, or positive cotinine test upon Screening or Check-in.
22. Receipt of blood products within 60 days prior to Check-in.
23. Donation of blood from 90 days prior to Screening, plasma from 14 days prior to Screening, or platelets from 42 days prior to Screening.
24. Poor peripheral venous access.
25. History of abnormal peripheral sensation including paraesthesia and/or numbness in arms and/or legs.
26. Have previously completed or withdrawn from this study or any other study investigating bevacizumab, and/or have previously received bevacizumab.
27. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects may be enrolled
Enrollment: 114 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunu Valasseri, MBBS, MSc, Principal Investigator — Covance; Muna Albayaty, MBChB,FFPM,MSc, Principal Investigator — Parexel
Locations (2):
- United Kingdom (2):
  - PAREXEL International - Northwick Park Hospital, Harrow
  - Covance Clinical Research Unit Limited, Leeds

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Started | 38 | 38 | 38
Completed | 38 | 37 | 38
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin® | Total
Number analyzed (Participants) | 38 | 38 | 38 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 38 | 114
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10.8) | 35 (9.1) | 38 (9.9) | 37 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 38 | 38 | 38 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 35 | 30 | 30 | 95
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 76.9 (9.38) | 77.9 (8.11) | 77.8 (8.29) | 77.6 (8.55)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (2.66) | 24.3 (2.61) | 25.0 (2.07) | 24.5 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Serum Concentration
Description: To compare the pharmacokinetic (PK) profiles of MB02, US Avastin® and EU Avastin® (in terms of Cmax) to establish bioequivalence between the 3 study arms.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) for the geometric LS means ratios are fully contained within the predefined bioequivalence limits of 0.80 to 1.25.
Time Frame: Predose, 1.5 h after end of infusion, 2, 3, 4, 5, 6, 8, 12, 24 h post-dose on Day 1-8, Day 10, Day 14, Day 21, Day 28, Day 42, Day 56, Day 78, and Day 100.
Population: Overall number of participants analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/(mg/mL)
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 38 | 38
(ng/mL)/(mg/mL) | 83000 (22.4) | 65200 (21.9) | 74400 (25.3)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (Cmax) falls completely within the range 0.80-1.25. The PK parameter Cmax was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.28, 90% CI 2-sided [1.18 to 1.39], Standard Deviation 0.05 — For the comparison, MB02 represents the numerator and US Avastin represents the denominator
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 1.12, 90% CI 2-sided [1.03 to 1.22], Standard Deviation 0.05 — For the comparison, MB02 represents the numerator and EU Avastin represents the denominator
Statistical Analysis 3: Comparison: US Licenced Avastin® vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 1.14, 90% CI 2-sided [1.05 to 1.24], Standard Deviation 0.05 — Ratio of GLSM, EU is the numerator and US Avastin acts as the denominator

2. Primary Outcome: AUC(0-∞); Area Under the Serum Concentration-time Curve From Time Zero to Infinity
Description: To compare the pharmacokinetic (PK) profiles of MB02, US Avastin® and EU Avastin® (in terms of AUC[0-∞]) to establish bioequivalence between the 3 study arms.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) for the geometric least square means (GLSM) ratios are fully contained within the predefined bioequivalence limits of 0.80 to 1.25.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
ng*h/mL | 28200000 (16.3) | 22900000 (17.8) | 24500000 (15.2)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 0.80-1.25. The PK parameter AUC[0-∞] was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.16, 90% CI 2-sided [1.09 to 1.22], Standard Deviation 0.05; For the comparison, MB02 represents the numerator and US Avastin represents the denominator
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.16, 90% CI 2-sided [1.09 to 1.22], Standard Deviation 0.05 — MB02 represents the numerator and EU Avastin represents the denominator
Statistical Analysis 3: Comparison: US Licenced Avastin® vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.07, 90% CI 2-sided [1 to 1.13], Standard Deviation 0.05 — EU Avastin corresponds to the numerator and US Avastin corresponds to the denominator

3. Secondary Outcome: Tmax: Time of Maximum Observed Serum Concentration
Description: To evaluate the tmax of MB02, US Avastin® and EU Avastin® .
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 38 | 38
h | 2.51 [1.62 to 71.98] | 4.00 [1.62 to 11.98] | 3.00 [1.57 to 12.00]

4. Secondary Outcome: AUC(0-t) = Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Observable Concentration;
Description: To evaluate the AUC[0-t] of MB02, US Avastin® and EU Avastin®.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
ng*h/mL | 27400000 (15.5) | 22300000 (16.9) | 23700000 (14.2)

5. Secondary Outcome: CL: Total Body Drug Clearance After IV Administration
Description: To evaluate the CL of MB02, US Avastin® and EU Avastin®
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: l/h
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
l/h | 0.00814 (16.5) | 0.0101 (17.9) | 0.00947 (15.4)

6. Secondary Outcome: t1/2: Apparent Serum Terminal Elimination Half-life
Description: To evaluate the t1/2 of MB02, US Avastin® and EU Avastin®
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
h | 451 (14.4) | 437 (15.5) | 449 (19.3)

7. Secondary Outcome: Immunogenicity
Description: Incidence of anti-bevacizumab antibodies (ADA), including neutralizing antibodies (Nab). Subjects who tested positive at baseline are not included here.
Time Frame: Day -1, Day 14, 28, 56, and 78
Measure: Count of Participants; unit: Participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 38 | 38
Participants
  ADA positive | 2 | 2 | 1
  nAb positive | 1 | 0 | 0
  NO seroconversion | 35 | 36 | 37

8. Secondary Outcome: Safety (Incidence of Treatment-related Adverse Events Using CTCAE v4.03)
Description: Compare the incidence of TEAEs reported in each treatment arm.
Time Frame: Day 1 - Day 100
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 38 | 38
participants
  Subjects with TEAEs | 24 | 28 | 25
  Subjects with SAEs | 0 | 1 | 0
  Subjects discontinued due to TEAEs | 0 | 0 | 0
  Related TEAEs | 6 | 3 | 8
  TEAEs of mild severity | 24 | 25 | 24
  TEAEs of moderate severity | 4 | 10 | 5
  TEAEs of severe severity | 0 | 1 | 0

9. Other Pre Specified Outcome: AUC(0-∞) Adjusted: Protein-adjusted Area Under the Serum Concentration-time Curve From Time Zero to Infinity
Description: Due to variability in the actual protein content between the study drugs and study drug batches which had the potential to influence the study results (as AUC is a dose-dependent PK parameter), protein-adjusted AUC(0-∞) was also derived for each individual by dividing each parameter by the actual protein content of the product batch that the individual subjects received.
  The 3 mg/kg IV dose of MB02 and US Avastin®, MB02 and EU Avastin®, and EU and US Avastin® were all considered bioequivalent in terms of the protein-adjusted AUCs and Cmax as the 90% CI for the geometric LS means ratios were fully contained within the predefined bioequivalence limits of 0.80 to 1.25 for all 3 comparisons. In general, as assessed from the geometric CV%, between-subject variability remained similar following protein adjustment compared to the unadjusted AUCs and Cmax.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
ng*h/mL | 1040000 (16.3) | 981000 (18.1) | 1020000 (14.5)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.02, 90% CI 2-sided [0.962 to 1.07], Standard Deviation 0.05 — MB02 in numerator and EU Avastin in denominator
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.06, 90% CI 2-sided [0.996 to 1.13], Standard Deviation 0.05 — MB02 is numerator and US Avastin is denominator
Statistical Analysis 3: Comparison: US Licenced Avastin® vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.04, 90% CI 2-sided [0.983 to 1.11], Standard Deviation 0.05 — EU Avastin in the numerator and US Avastin in the denominator

10. Other Pre Specified Outcome: AUC(0-t) Adjusted: Protein Adjusted Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Observable Concentration
Description: Due to variability in the actual protein content between the study drugs and study drug batches which had the potential to influence the study results (as AUC is a dose-dependent PK parameters), protein-adjusted AUC(0-t) was also derived for each individual by dividing each parameter by the actual protein content of the product batch that the individual subjects received.
  The 3 mg/kg IV dose of MB02 and US Avastin®, MB02 and EU Avastin®, and EU and US Avastin® were all considered bioequivalent in terms of the protein-adjusted AUCs and Cmax as the 90% CI for the geometric LS means ratios were fully contained within the predefined bioequivalence limits of 0.80 to 1.25 for all 3 comparisons. In general, as assessed from the geometric CV%, between-subject variability remained similar following protein adjustment compared to the unadjusted AUCs and Cmax.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 37 | 38
ng*h/mL | 1010000 (15.5) | 955000 (17.2) | 991000 (13.6)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.02, 90% CI 2-sided [0.969 to 1.07], Standard Deviation 0.05 — MB02: EU Avastin
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.06, 90% CI 2-sided [0.998 to 1.12], Standard Deviation 0.05 — MB02: US Avastin
Statistical Analysis 3: Comparison: US Licenced Avastin® vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.04, 90% CI 2-sided [0.981 to 1.1], Standard Deviation 0.05 — EU Avastin: US Avastin

11. Other Pre Specified Outcome: Cmax Adjusted: Protein Adjusted Maximum Observed Serum Concentration
Description: Due to variability in the actual protein content between the study drugs and study drug batches which had the potential to influence the study results (as Cmax is a dose-dependent PK parameters), protein-adjusted Cmax was also derived for each individual by dividing each parameter by the actual protein content of the product batch that the individual subjects received.
  The 3 mg/kg IV dose of MB02 and US Avastin®, MB02 and EU Avastin®, and EU and US Avastin® were all considered bioequivalent in terms of the protein-adjusted AUCs and Cmax as the 90% CI for the geometric LS means ratios were fully contained within the predefined bioequivalence limits of 0.80 to 1.25 for all 3 comparisons. In general, as assessed from the geometric CV%, between-subject variability remained similar following protein adjustment compared to the unadjusted AUCs and Cmax.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/(mg/mL)
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
Number analyzed (Participants) | 38 | 38 | 38
(ng/mL)/(mg/mL) | 3050 (22.4) | 2790 (22.1) | 3110 (25.2)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 0.986, 90% CI 2-sided [0.903 to 1.08], Standard Deviation 0.05 — MB02: EU Avastin
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.1, 90% CI 2-sided [1.01 to 1.19], Standard Deviation 0.05 — MB02: US Avastin
Statistical Analysis 3: Comparison: US Licenced Avastin® vs EU Approved Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 1.12, 90% CI 2-sided [1.02 to 1.22], Standard Deviation 0.05 — EU Avastin: US Avastin

ADVERSE EVENTS:
Time Frame: Study duration (Day 1 - Day 100)
Description: Coded according to Medical Dictionary for Regulatory Activities (version 20.1), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 4.03).
  Following a request from the Medicines and Healthcare products Regulatory Authority (MHRA) all serious adverse reactions were considered unexpected and reported as SUSARs, for the purpose of safety reporting in healthy volunteers.
Arm/Group | MB02 (Bevacizumab Biosimilar) | US Licenced Avastin® | EU Approved Avastin®
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/38 | 0/38
Other Adverse Events (participants affected / at risk) | 24/38 | 28/38 | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB02 (Bevacizumab Biosimilar) (N=38) | US Licenced Avastin® (N=38) | EU Approved Avastin® (N=38)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB02 (Bevacizumab Biosimilar) (N=38) | US Licenced Avastin® (N=38) | EU Approved Avastin® (N=38)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (9) | 8 (10) | 8 (10)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (5) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 11 (12) | 6 (7)
Nasophyringitis (Infections and infestations) | 2 (2) | 4 (6) | 5 (6)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03293654/Prot_004.pdf
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03293654/SAP_005.pdf